CLINICAL TRIAL: NCT02950012
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Study to Evaluate the Efficacy and Safety of OPTI-BIOME™ Bacillus Subtilis MB40 on Abdominal Discomfort, Gas and Bloating in a Healthy Population
Brief Title: A Study to Evaluate OPTI-BIOME™ Bacillus Subtilis MB40 on Abdominal Discomfort, Gas and Bloating in a Healthy Population
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BIO-CAT Microbials, LLC (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Organization: BIO-CAT, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 16OBHB
Record Dates: First submitted 2016-10-28; First posted 2016-10-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Bloating
Keywords: Healthy; Bloating; Abdominal Discomfort; Gas; Probiotic; Bacillus Subtillis
MeSH Terms: conditions — Mucopolysaccharidosis IV

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OPTI-BIOME™ Bacillus subtilis MB40 (Experimental)
  Interventions: Dietary Supplement: OPTI-BIOME™ Bacillus subtilis MB40
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: OPTI-BIOME™ Bacillus subtilis MB40
  Arms: OPTI-BIOME™ Bacillus subtilis MB40
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effects of OPTI-BIOME™ (Bacillus subtilis MB40), a probiotic supplement, on bloating, gas and abdominal discomfort symptoms in otherwise healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18-75 years (inclusive) of age
2. BMI 18.5-29.9 ±1 kg/m2
3. Abdominal bloating intensity score ≥5 and at least two days of bloating over the 2 weeks prior to screening (assessed at screening by Abdominal Bloating questionnaire)
4. Participants categorized as 'high bloaters' as defined by an average bloating score ≥ 5 during the run-in period assessed at baseline by question 3 of the Modified Daily Abdominal Discomfort, Gas, and Bloating Questionnaire, AND/OR, participants categorized as 'high frequency bloaters' as defined by greater than 7 days of high bloating (defined above) during the run-in period.

   * For females, this should not include abdominal discomfort or bloating experienced during menstruation, if such symptoms occur due to menstrual cycle females should go through another run-in period.
5. If female, participant is not of child bearing potential, which is defined as females who have had a hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation) OR

   Females of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result. Acceptable methods of birth control include:
   * Hormonal contraceptives (stable for 1 month) including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner (shown successful as per appropriate follow-up)
6. Healthy as determined by laboratory results, medical history, and physical exam
7. Agrees to abstain from consuming unpasteurized bacteria-fermented foods including cheese and yogurt for 1 week prior to screening visit and throughout the study
8. Agrees to abstain from using fiber supplements 2 weeks prior to screening and for the duration of the study
9. Agrees to maintain current dietary habits and activity/training levels for two weeks prior to baseline and for the course of the study
10. Agrees to avoid probiotics for one week prior to screening and for the course of the study
11. Willingness to complete all the study requirements and attend all clinic visits.
12. Has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

1. Females who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial
2. History of chronic inflammation or structural abnormality of the digestive tract (inflammatory bowel disease, duodenal or gastric ulcer, intestinal obstruction, or symptomatic cholelithiasis)
3. Nocturnal and/or progressive abdominal pain (abdominal pain that increases in intensity and is consistent on regular basis)
4. Significant weight loss over the past 3 months (significance to be determined by the Qualified Investigator)
5. Type 1 and type 2 diabetes
6. History of colorectal cancer, anal abscess, anal fistula, anal fissure, anal stenosis, gastric retention or obstruction, bowel resection, rectocele, or colostomy
7. Cancer except skin cancers completed excised with no chemotherapy or radiation following and with a negative follow up.
8. Diagnosis of adenomatous polyposis, irritable bowel syndrome, chronic gastritis or functional dyspepsia, crohn disease, and celiac disease Renal or hepatic insufficiency
9. Gastrointestinal bleeding or acute infection
10. Immunodeficiency
11. History of organ transplant
12. Use of antibiotics within 4 weeks of randomization Routine (at least 3 times per week) consumption of probiotic or prebiotic supplements or supplemented foods and are unwilling to stop at least one week prior to screening and throughout the study
13. Use of immunosuppressant drugs
14. Change in anti-psychotic medication within 3 months of randomization
15. Abdominal surgery within 6 months of randomization
16. Plan to donate blood during the study or within 30 days of completing the study
17. Participation in a clinical research trial within 30 days prior to randomization
18. Allergy or sensitivity to study supplement or placebo ingredients
19. Alcohol abuse (>2 standard alcoholic drinks per day) or drug abuse within the last 6 months
20. Use of Medicinal Marijuana
21. Cognitively impaired and/or unable to give informed consent
22. Unstable medical conditions
23. Clinically significant abnormal laboratory results at screening
24. Any other condition which in the Qualified Investigator's opinion may adversely affect the volunteer's ability to complete the study or its measures or which may pose significant risk to the volunteer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-10; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Weekly mean of the daily bloating scores | 4 weeks
  Discomfort, Gas and Bloating questionnaire

SECONDARY OUTCOMES:
Weekly mean of the daily gas score (flatulence) | 4 weeks
  Discomfort, Gas and Bloating questionnaire
Weekly mean of the abdominal pain score | 4 weeks
  Discomfort, Gas and Bloating questionnaire
Modified Gastrointestinal Symptom Rating Scale (GSRS) score | 4 weeks
Weekly mean stool consistency scores | 4 weeks
  Bristol stool scale
Weekly mean number of bowel movements | 4 weeks
  Daily Bowel Habits Diary
Quality of Life | 4 weeks
  Rand SF-36

OTHER OUTCOMES:
Incidence of clinically significant abnormal vital signs | 4 weeks
Incidence of clinically significant abnormal complete blood panel | 4 weeks
Incidence of clinically significant abnormal electrolytes | 4 weeks
Incidence of clinically significant abnormal kidney function panel | 4 weeks
Incidence of clinically significant abnormal liver function panel | 4 weeks
Incidence of adverse events | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tetyana Pelipyagina, MD', Principal Investigator — KGK Science Inc.
Locations (3):
- United States (2):
  - KGK Clinical Trials Center, Foothill Ranch, California
  - KGK Clinical Trials Center, Orlando, Florida
- KGK Synergize Inc., London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Penet C, Kramer R, Little R, Spears JL, Parker J, Iyer JK, Guthrie N, Evans M. A Randomized, Double-blind, Placebo-controlled, Parallel Study Evaluating the Efficacy of Bacillus subtilis MB40 to Reduce Abdominal Discomfort, Gas, and Bloating. Altern Ther Health Med. 2021 Jun;27(S1):146-157. PMID 31719214